CLINICAL TRIAL: NCT00262990
Title: A Randomized, Parallel Group, Open-label, Active Controlled, Multicenter Phase III Trial of Patupilone (EPO906) Versus Pegylated Liposomal Doxorubicin in Taxane/Platinum Refractory/Resistant Patients With Recurrent Epithelial Ovarian, Primary Fallopian or Primary Peritoneal Cancer
Brief Title: Patupilone Versus Doxorubicin in Patients With Ovarian, Primary Fallopian, or Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2303
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-05

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Neoplasms
Keywords: Epithelial ovarian cancer; fallopian tube cancer; peritoneal cancer; primary cancer; recurrent cancer; doxorubicin; taxane chemotherapy; platinum chemotherapy; Patupilone; taxane platinum resistant
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Carcinoma, Ovarian Epithelial; Neoplasms; Recurrence | interventions — epothilone B; Doxorubicin

ARMS (2):
- Patupilone (Experimental)
  Interventions: Drug: EPO906 (Patupilone)
- doxorubicin (Active Comparator)
  Interventions: Drug: doxorubicin

INTERVENTIONS:
Drug: EPO906 (Patupilone)
  Other Names: Patupilone
  Arms: Patupilone
Drug: doxorubicin
  Arms: doxorubicin

SUMMARY:
The objective of this study is to assess the safety and efficacy of patupilone compared to pegylated liposomal doxorubicin. Additionally, this study will assess the ability of patupilone to extend the survival time and potential beneficial effects in women who have nonresponsive or recurrent ovarian, primary fallopian, or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Confirmed diagnosis of ovarian, fallopian or peritoneal cancer
* No more than three chemotherapy regimens
* Most recent regimen must have been platinum based

Exclusion Criteria:

* Have an unresolved bowel obstruction
* Have had previous chemotherapy within 3 weeks
* Recovering from any surgery for any cause

Other protocol-defined inclusion/exclusion criteria will apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2005-11; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To show superiority of patupilone in overall survival compared to doxorubicin in taxane/platinum resistant patients with ovarian cancer | every 8 weeks

SECONDARY OUTCOMES:
To determine the duration of overall response in patients with complete response (CR) or partial response (PR) or stable disease (SD) | End of study
To determine the progression-free survival (PFS) of patients treated with patupilone | end of study
To determine the time to disease progression (TTP) of patients treated with patupilone | end of study
To determine overall best tumor response (CR, PR, SD, PD and Unknown) | end of study
To investigate the safety and tolerability of patupilone | end of study
To evaluate the pharmacokinetics (PK) of patupilone from all patients | end of study
To explore relationships between Cmin (pre-dose patupilone blood concentration) and efficacy/adverse events | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (148):
- United States (103):
  - Alaska Cancer Research & Education Center, Anchorage, Alaska
  - Northern Arizona Hematology & Oncology Associates, Flagstaff, Arizona
  - Mayo Center for Women's Health, Scottsdale, Arizona
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Yanagihara, Ronald H., Gilroy, California
  - California Cancer Care, Inc., Greenbrae, California
  - University of California - San Diego/ Moores Cancer Center, La Jolla, California
  - LAC & USC Women's & Children's Hospital, Los Angeles, California
  - Gynecologic Oncology associates, Newport Beach, California
  - UC Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - Anschutz Cancer Pavilion - Clinical Investigations Core, Aurora, Colorado
  - University Of Colorado Health Sciences Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Gynecologic Oncology, LLC, Newark, Delaware
  - Washington Hospital Center/Medstar Research Institute, Washington D.C., District of Columbia
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Miami Cancer Center at Mercy Hospital, Miami, Florida
  - Miami Cancer Center at University Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Mt. Sinai Medical Center, Miami, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - MD Anderson Cancer Center of Orlando, Orlando, Florida
  - Oncology & Hematology Associates of West Broward, Tamarac, Florida
  - Xelero Medical Research/Giselle Ghurani, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children/Univ. of HI, Honolulu, Hawaii
  - Northwest Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Institute of Central Illinois/Decatur Memorial Hospital, Decatur, Illinois
  - Indiana University Obstetrics, Indianapolis, Indiana
  - Indiana University Cancer Center/Indiana UNiversity Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - Gynecologic Oncology of Indiana/St. Francis Cancer Research Foundation, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Louisville Oncology, Louisville, Kentucky
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Boston University Medical Center Hospital, Boston, Massachusetts
  - Providence Cancer Center, Southfield, Michigan
  - Minnesota Oncology/Hematology, PA, Burnsville, Minnesota
  - St. Luke's Hospital, Duluth, Minnesota
  - Minnesota Oncology/Hematology, PA, Edina, Minnesota
  - Minnesota Oncology/Hematology Associates of Central Illinois, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Metro-MN CCOP, Saint Louis Park, Minnesota
  - Minnesota Oncology Hematology, Saint Paul, Minnesota
  - The West Clinic, Corinth, Mississippi
  - The West Clinic, Southaven, Mississippi
  - St. Luke's Hospital of Kansas City/St. Luke's Cancer Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Southeast Nebraska Oncology/Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hematology and Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - University of Medicine and Dentistry of New Jersey/The Cancer Institute of Neew Jersey, New Brunswick, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Schwartz Gynecologic Oncology, PLLC, Babylon, New York
  - Bellview Hospital, New York, New York
  - New York University School of Medicine/NYU Cancer Institute, New York, New York
  - NYU Cancer Institute, New York, New York
  - St. Vincent Catholic Medical Center of New York, Staten Island, New York
  - Brody School of Medicine, Greenville, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Camelot Women's Cancer, Columbus, Ohio
  - The Arthur G. James Cancer Hospital, Columbus, Ohio
  - Cancer Care Associates, Tulsa, Oklahoma
  - Oncology Associates of Oregon, PC/Willaimette Valley Cancer Center, Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Willamette Valley Cancer Center, Springfield, Oregon
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - Magee - Women's Hospital, Pittsburgh, Pennsylvania
  - GYN Oncology Research/Gynecologic Oncology Research & Development, LLC, Greenville, South Carolina
  - Chattanooga GYN Oncology, Chattanooga, Tennessee
  - Hall and Martin MDs, PC, Knoxville, Tennessee
  - The West Clinic, Memphis, Tennessee
  - West Clinic, Memphis, Tennessee
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology, Austin, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Oncology Consultants P.A., Houston, Texas
  - Cancer Care Center of South Texas, San Antonio, Texas
  - Waco Cancer Care & Research Center, Waco, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - Cancer Outreach Associates, Abingdon, Virginia
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University/VCU Massey Cancer Center, Richmond, Virginia
  - Gersh, Robert, Spokane, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Aurora Medical Gyn Group, West Allis, Wisconsin
- Australia (6):
  - Novartis Investigative Site, Adelaide
  - Novartis Investigative Site, Herston
  - Novartis Investigative Site, Nedlands, WA
  - Novartis Investigative Site, South Brisbane
  - Novartis Investigative Site, St Leonards
  - Novartis Investigative Site, Wodonga
- Canada (7):
  - BC Cancer Agency, Vancouver, British Columbia
  - Novartis Investigative Site, Calgary
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, North York
  - Novartis Investigative Site, Québec
  - Novartis Investigative Site, Sherbrooke
  - Novartis Investigative Site, Toronto
- Denmark (2):
  - Novartis Investigative Site, Odense
  - Novartis Investigative Site, Vejle
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Tampere
- France (5):
  - Novartis Investigative Site, Amboise
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Herblain Cedec
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Athens, Greece
- Italy (7):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Monza
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Torino
- Novartis Investigative Site, Krakow, Poland
- South Africa (7):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Johannesburg, Gauteng
  - Novartis Investigative Site, Klerksdorp
  - Novartis Investigative Site, Port Elizabeth
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Pretoria, Guateng
  - Novartis Investigative Site, Sandton, Gauteng
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- United Kingdom (4):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Metropolitan Borough of Wirral
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Colombo N, Kutarska E, Dimopoulos M, Bae DS, Rzepka-Gorska I, Bidzinski M, Scambia G, Engelholm SA, Joly F, Weber D, El-Hashimy M, Li J, Souami F, Wing P, Engelholm S, Bamias A, Schwartz P. Randomized, open-label, phase III study comparing patupilone (EPO906) with pegylated liposomal doxorubicin in platinum-refractory or -resistant patients with recurrent epithelial ovarian, primary fallopian tube, or primary peritoneal cancer. J Clin Oncol. 2012 Nov 1;30(31):3841-7. doi: 10.1200/JCO.2011.38.8082. Epub 2012 Sep 17. PMID 22987083
- See also: In the search box enter NCT00262990 — http://www.clinicaltrials.gov
- See also: Select "Ovarian Cancer" — http://www.novartisclinicaltrials.com
- See also: Results for CEPO906A2303 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3944